CLINICAL TRIAL: NCT03596957
Title: Subacute Effect of Tolvaptan on Total Kidney Volume in Adult Patients With Autosomal Dominant Polycystic Kidney Disease
Acronym: PoCKET
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lisbet Brandi (Other)
Responsible Party: Sponsor-Investigator, Lisbet Brandi, Head of Department for Endrocrinology and Nephrology, MD, DMSc, MHM, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PoCKET
Record Dates: First submitted 2018-02-14; First posted 2018-07-24 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Autosomal Dominant Polycystic Kidney
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Intervention Model Description: Patients will be randomised in a 1:1 ration either to treatment with tolvaptan for six weeks followed by six weeks observation without trial medicaion or to the Control group receiving no tolvaptan treatment for 12 weeks
Who Masked: Outcomes Assessor
Masking Description: The endpoint blinding will be assured since all the MRI scans will be forwarded to the Comparative Medicine Laboratory in Aarhus for evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tolvaptan group (Active Comparator): Treatment with tolvaptan for six weeks followed by six weeks observation without trial medication
  Interventions: Drug: Tolvaptan
- Control group (No Intervention): No tolvaptan treatment but following the same visit and investigation plan as the subjects in the tolvaptan group

INTERVENTIONS:
Drug: Tolvaptan — At baseline the tolvaptan dosing will start with daily morning and afternoon doses of 45 mg and 15 mg respectively, with weekly increases to 60 mg and 30 mg and then to 90 mg and 30 mg according to subject tolerability
  Other Names: Jinarc
  Arms: Tolvaptan group

SUMMARY:
Investigator initiated controlled multi-centre trial in a Prospective, Randomised, Open, Blinded Endpoint (PROBE) design.

Patients will be randomised in a 1:1 ratio either to treatment with tolvaptan for six weeks followed by six weeks observation without trial medication or no tolvaptan treatment, but following the same visit and investigation plan as the subjects taking tolvaptan.

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) is the most common genetic kidney disease and the fourth leading cause of end-stage renal disease in adults Worldwide.

The tolvaptan tablet has been approved by EMA (European Medicines Agency) with the indication of slowing the progression of cysts development and renal insufficiency in adults with ADPKD. It is the newest and only possible treatment for this patient group and could be initiated in patients with evidence for rapidly progressive disease Development.

There is however in Denmark and other countries both scientific and financial reluctance to initiate this expensive treatment for several reasons e.g. selection of patients who might benefit, effect on progression of kidney disease, side effects and tolerability.

Before deciding on implementation in Denmark, more knowledge is needed. The results of the PoCKET trial will contribute with guidance on this decision.

Foremost the trial is designed to address not only the change in kidney volume, but the change in kidney function, which is what matters to the patients and their prognosis in terms of postponing time to end stage renal disease. Furthermore, important data on side effects and tolerability will be generated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18 and 65 years
* Diagnosis of typical ADPKD
* tKV above or equal to 750 ml by MRI scanning
* Estimated GFR (e-GFR) by CKD-EPI formula of above or equal to 45 mL/min/1.73 m2

Exclusion Criteria:

* Kidney transplant recipient
* Known liver disease except for liver cysts relating to ADPKD
* ASAT and ALAT above upper normal level
* Current treatment with thiazide and thiazide-line diuretics, mineral corticoid receptor antagonists, amiloride or loop diuretics
* Evidence of urinary tract obstruction
* Current treatment with CYP3A4 inhibitors
* Active malignant disease
* Current or previous treatment with tolvaptan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in total Kidney Volume (tKV) measured by MRI scanning | Between baseline and six weeks and between six and 12 weeks
  The change in the total Kidney Volume after six and 12 weeks participation in the trial

SECONDARY OUTCOMES:
Changes in GFR | Between baseline and six weeks and between baseline and 12 weeks
  The changes in GFR measured by Cr-EDTA clearance
Changes in relevant genetic and non-genetic biomarkers associated with CKD and ESRD | Between baseline and six weeks and between baseline and 12 weeks
  Prediction of change in progression of the disease over time in the genes PKD1, PKD2, PKHD1 and HNF1B. The following biomarkers will be determined: NGAL, UMOD, MCP-1, KIM-1, cystatin-C and copeptin
Changes in Quality of Life | Between baseline and six weeks and between baseline and 12 weeks
  Questionnaire SF36 Health Survey - with 36 questions to subject's health and wellbeing
Subject estimation of own health | Between baseline and six weeks and between baseline and 12 weeks
  Estimated by a Visual Analogue Scale from 0 (worth wellbeing) to 100 (best wellbeing
Changes in ASAT and ALAT | Between baseline and six weeks and between baseline and 12 weeks
  Changes estimated from laboratory results
Incidence of Adverse Events | Between baseline and six weeks and between baseline and 12 weeks
  Evaluation of Adverse Events including severity, causality, outcome and seriousness assessments

CONTACTS AND LOCATIONS:
Overall Officials: Lisbet Brandi, MD DMSc MHM, Principal Investigator — KNEA, Nordsjaellands Hospital
Locations (6):
- Denmark (6):
  - Aarhus University Hospital - Site 43, Skejby, Aarhus N
  - Odense University Hospital - Site 45, Odense, Odense C
  - Rigshospitalet - Site 42, Copenhagen
  - Herlev Hospital, Herlev
  - Nordsjaellands Hospital - Site 41, Hillerød
  - Sjællands University Hospital Roskilde, Roskilde